CLINICAL TRIAL: NCT03310762
Title: The Effect of Using Vaccine Reminder and Tracker Bracelets to Improve Routine Childhood Immunization Coverage and Timeliness in Pakistan: a Randomized Control Trial.
Brief Title: Immunization Reminder Bracelets Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Interactive Research and Development (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Danya Arif, Program Manager, Interactive Research and Development
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 027562-746846- 0303
Record Dates: First submitted 2017-09-22; First posted 2017-10-16 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Immunization; Infection
Keywords: immunization coverage; silicon bracelet; immunization reminders
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: This is an individually randomized, three-arm parallel group design randomized control trial with equal allocation in the two treatment groups and control group. Children in intervention group A will receive the simple silicon bracelets, children in intervention group B will receive the bracelets developed by Alma Sana Inc. and children in the Control group will not receive any intervention.
Masking Description: The allocation sequence will be concealed from the study staff responsible for screening and enrolling participants in serially numbered, opaque, sealed envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alma Sana Bracelet Arm (Experimental): Subjects in this arm will receive a vaccine reminder and tracker bracelet developed by Alma Sana Inc. This bracelet uses a combination of symbols and numbers to denote the entire vaccine schedule a child is supposed to receive before the age of 2 years. Shapes indicate vaccines, and numbers signify the child's age.
  Interventions: Other: Alma Sana Bracelet
- Simple Silicon Bracelet Arm (Experimental): Subjects in this arm will receive a simple silicon bracelet. This bracelet has six symbols to remind parents that their child needs to get at least six vaccination visits before he reaches 2 years of age. The first five symbols are represented by a crescent shape and the sixth symbol is represented by a star shape to denote that the child is fully immunized.
  Interventions: Other: Simple Silicon Bracelet
- Control Arm (No Intervention): Subjects in this arm will not receive any bracelet/intervention.

INTERVENTIONS:
Other: Alma Sana Bracelet — Every time a child receives a vaccine, vaccinators will hole punchers to perforate shapes denoting the particular vaccine a child has received.
  Arms: Alma Sana Bracelet Arm
Other: Simple Silicon Bracelet — Every time a child receives a vaccine, vaccinators will hole punchers to perforate shapes denoting the particular vaccine a child has received.
  Arms: Simple Silicon Bracelet Arm

SUMMARY:
Pakistan has one of the highest infant mortality rates in the world in part, due to the low coverage (54%) for all basic vaccinations. Low uptake, lack of awareness among parents to complete the recommended immunization schedule and inability to remember vaccine appointments are some of the key factors hindering improvement in uptake of immunization services. On the supply side, ineffective methods to track children's' vaccine doses means that there is no reliable mechanism to verify vaccine administration and estimate accurate immunization coverage.

This study proposes to develop and test two types of silicon bracelets for children to stimulate immunization demand and simultaneously address supply side verification issues. These bracelets use a combination of numbers and symbols to denote the age of the child and due vaccines and are designed for illiterate or uneducated mothers; are low-cost and adaptable to most local settings. At the time of vaccine administration, the appropriate symbol denoting the vaccine on the bracelets is punched and therefore the bracelets can serve as effective reminders for mothers for timely immunization of their child and as a tool for vaccinators to verify vaccine administration and coverage.

An individually randomized, three-arm parallel group design randomized control trial will be conducted with equal allocation in the two treatment groups and control group. Children in intervention group A will receive the simple silicon bracelets, children in intervention group B will receive the bracelets developed by Alma Sana Inc. and children in the Control group will not receive any intervention. The impact of these immunization reminder bracelets on immunization coverage and timeliness will be evaluated through a randomized control trial (RCT) across 4 immunization centers in Karachi. To evaluate the bracelets' impact, variables of interest-coverage and timeliness rates of pentavalent-3/PCV-3/polio-3 and Measles 1 vaccine will be compared between Group A and the Control Group and Group B and the Control Group.

Proposed results include increase in immunization coverage and timeliness of Pentavalent-3/Pneumococcal Conjugate Vaccine (PCV-3)/Polio-3 and Measles-1 in the intervention versus control group.

The study will provide evidence of the bracelet's effectiveness for the global health community and provide a simple tool for strengthening routine immunization efforts in Pakistan.

DETAILED DESCRIPTION:
The overall goal of the intervention is improvement in both immunization coverage rates and timeliness among the study participants through introducing simple silicon bracelets as childhood vaccination reminders and trackers.

An individually randomized, three-arm parallel group design randomized control trial will be conducted with equal allocation to evaluate the impact of the Alma Sana bracelet and simple silicon bracelet by comparing the variables of interest (coverage and timeliness rates of (pentavalent-3/PCV-3/polio-3 and Measles 1) between treatment groups and the Control Group.

Study Procedures:

A consent form will be used to seek consent from caregivers accompanying the child to screen the child for the study. Among those who provide consent, a screening form will be used to identify the eligible participants. After screening, seeking consent from primary caregivers (mother and/or father) they will be randomized into the treatment groups (to receive the bracelet) or to serve as a control. The randomization sequence will be created using Stata version 13 with a 1:1:1 allocation using random block sizes of 3, 6, 9 and 12. The allocation sequence will be concealed from the study staff responsible for screening and enrolling participants in serially numbered, opaque, sealed envelopes. After randomization, each child will be assigned a unique study ID (a sticker containing the study ID will be pasted on the child's government issued EPI card).

Details of the procedures in the intervention and control groups are outlined below:

Intervention group A and B: Children in both the intervention groups (A and B) will receive the two different bracelets to be placed on the child's wrist. Additionally, mothers will be provided instructions explaining the use of the bracelet and helping them decode the symbols to enable them to use the bracelet to remind themselves of their child's vaccinations. Children will receive the scheduled EPI vaccine by the vaccinator who will then punch a hole in the child's bracelet to denote vaccine administration. The child's vaccine data will be recorded in the EPI card and EPI register as per routine.

All participants (irrespective of whether they are in the treatment group A or B or control group) will receive the routine EPI vaccinations as per Pakistan's EPI Immunization schedule (one dose of BCG and polio soon after birth, 3 doses of Pentavalent/Polio/PCV at 6, 10 and 14 weeks, and 2 doses of Measles vaccine and 9 and 15 months of age) and the vaccinator will record the child's immunization data in the EPI immunization card as well as EPI register. The difference between the intervention and standard care is only the provision of bracelets which provide an additional source (apart from the EPI cards) to record and track vaccinations.

Control group: Children in the control group will receive the scheduled EPI vaccine from the vaccinator. The child's vaccine data will be recorded in the EPI card and register as per routine.

Data collection will be done using the following documents over 5 total visits:

1. Enrollment Form: At the child's first visit to the center, the field worker will note the name and age of the child along with the immunizations received during the visit in addition to basic demographic information in the enrolment form. This information, along with basic biographic information is recorded routinely by vaccinators in their government issued permanent medical registers. An immunization visit typically takes between 10 and 15 minutes, not including any time spent waiting to be seen by the vaccinator.
2. Follow-up Form: For the follow up visits by the caregivers to get the subsequent vaccinations (3 - 4 visits), field workers will be based at the participating EPI centers throughout the follow-up period. Each follow-up visit takes about 10-15 minutes of the caregivers time, not including any time spent waiting to be seen by the vaccinator. Each child in the study is provided a unique EPI number by the EPI staff as per routine and also a study ID by a field worker. The linkage between the EPI number and the ID number will be maintained after data collection is complete. The field workers will use these IDs to identify the study participants when they come for follow-up visits. At each follow up visit, the field worker will record the vaccine administered and date for each child in the study, including verifying data on past immunizations and due vaccines (follow-up form attached). Therefore, for each study participant, the field workers would collect data 3-4 times during the follow-up period. The minimum duration of follow up provided to each participant will be until the child receives Measles-1 vaccine (given at 9 months of age per WHO recommendations). The maximum duration of follow up provided to each participant will be 11 months.
3. Completion Form: After the completion of follow-up period, short (15-20 minutes) phone or in-person interviews will be conducted to collect follow up vaccination data (if missing) and data on experiences of study participants regarding the bracelets (completion form attached). Phone numbers and addresses are provided as part of the Enrollment form. It is culturally acceptable for in person interviews to be conducted in their home. Key data points would include reasons for drop-outs, whether mothers understood how to use the bracelets, how often mothers said their babies wore the bracelets and why, what mothers liked and disliked about the bracelets and whether mothers would continue using the bracelets as reminders moving forward.

Statistical analysis plan:

Intention to treat analysis will be used-that is, all subjects will be analysed with the assumption that they remained in the treatment group to which they were initially assigned.

Y=c+β1T1+β2T2+γX+ε

Y is the relevant outcome measure (for instance Penta-3 coverage) C is the constant that gives the value of the outcome for the control group T1 and T2 are treatment dummy variables for group 1 (Alma Sana bracelets) and group 2 (Simple silicon bracelets) β1 and β2 will provide the difference in outcome variable between treatment one and the control group and treatment 2 and the control group respectively X is the set of possible covariates (gender, mother's education)

Logistic regression will be used to determine whether the difference in outcome between the two treatment groups and control group are statistically significant and whether the difference in outcome between the two treatment groups is statistically significant from each other.

ELIGIBILITY:
Inclusion Criteria:

1. Child is visiting the center for BCG or Pentavalent-1/Polio-1/PCV-1 vaccination.
2. Child is healthy
3. Child's caregiver has been a resident of study area for more than 6 months
4. Child is accompanied by a primary caregiver (mother and/or father)

Exclusion Criteria:

1. Child's age is more than 3 months. The average age of children for Penta-1 vaccine visit in Pakistan is 2.2 months (approximately 10 weeks). Children older than 3 weeks will be excluded on account of exceeding the average age for Penta-1 administration.
2. Parents plan to go to a different center for completing the vaccination course

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1445 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Increase in immunization coverage in intervention versus control | The outcome will be measured after at least 9 months of follow up of the last participant enrolled
  The primary outcome measure is the increase in coverage (i.e. the proportion of children getting vaccinated for) Pentavalent-3/PCV-3/polio-3 and Measles 1 vaccine in intervention versus control arm.
Increase in timeliness of immunization in intervention versus control | The outcome will be measured after at least 9 months of follow up of the last participant enrolled
  The primary outcome measure is the increase in timeliness of Pentavalent-3/PCV-3/polio-3 and Measles 1 vaccine in intervention versus control arm. Timeliness is defined as the proportion of children getting vaccinated for a particular antigen within the specified time duration i.e. a timely dose of Pentavalent-3/PCV-3/polio-3 is administered when the child is between 14 weeks and 22 weeks of age.

SECONDARY OUTCOMES:
Comparison of timely immunization coverage rates between treatment groups | The outcome will be measured after at least 9 months of follow up of the last participant enrolled
  Compare the proportion of children receiving timely doses of Pentavalent-3/PCV-3/polio-3 and Measles 1 vaccine in the Alma Sana group and the simple silicon bracelets group.

CONTACTS AND LOCATIONS:
Overall Officials: Danya A Siddiqi, MSc, Principal Investigator — Interactive Research and Development
Locations (4):
- Pakistan (4):
  - Future Colony, Karachi, Sindh
  - KMC Maternity Home, Karachi, Sindh
  - MCH-36B, Karachi, Sindh
  - Urban Health Center, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siddiqi DA, Ali RF, Munir M, Shah MT, Khan AJ, Chandir S. Effect of vaccine reminder and tracker bracelets on routine childhood immunization coverage and timeliness in urban Pakistan (2017-18): a randomized controlled trial. BMC Public Health. 2020 Jul 11;20(1):1086. doi: 10.1186/s12889-020-09088-4. PMID 32652969
- [Derived] Siddiqi DA, Munir M, Shah MT, Khan AJ, Chandir S. Effect of vaccine reminder and tracker bracelets on routine childhood immunization coverage and timeliness in urban Pakistan: protocol for a randomized controlled trial. BMC Public Health. 2019 Oct 30;19(1):1421. doi: 10.1186/s12889-019-7667-3. PMID 31666039